CLINICAL TRIAL: NCT03948789
Title: Multicenter, Randomized Phase III Study of MR-Guided Focused Ultrasound Surgery for the Treatment of Uterine Fibroids (MRgFUS TUF) Compared to Myomectomy in Symptomatic Medication and Not Sufficiently Treatable Uterine Fibroids
Brief Title: Phase III Study of MR-Guided Focused Ultrasound Surgery for the Treatment of Uterine Fibroids Compared to Myomectomy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARGI-T
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Myomectomy; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A Myomectomy (Active Comparator): Removement of uterine fibroids by myomectomy
  Interventions: Procedure: Myomectomy (laparoscopic or open surgical)
- B MRgFUS-TUF (Experimental): Removement of uterine fibroids by Magnetic Resonance Imaging-controlled high-focussed ultrasound therapy (MRgFUS-TUF)
  Interventions: Procedure: Magnetic Resonance Imaging-controlled high-focussed ultrasound therapy

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging-controlled high-focussed ultrasound therapy — Magnetic Resonance Imaging-controlled high-focussed ultrasound
  Arms: B MRgFUS-TUF
Procedure: Myomectomy (laparoscopic or open surgical) — Myomectomy (laparoscopic or open surgical)
  Arms: A Myomectomy

SUMMARY:
The aim of the study is to answer the question, whether in patients with symptomatic and medically not sufficiently treatable uterine fibroids (population) the "Magnetic-Resonance-Guided Focused Ultrasound Surgery" short, MRgFUS-TUF (intervention) offers less burdensome therapy and patient-relevant advantages (symptom relief) compared to the operative myomectomy (comparison). The study will hence investigate the therapeutic benefit of this method.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic and medically untreatable uterine fibroids who score at least 40 points on the Symptom Severity Score (SSS) of the Uterine Fibroid Symptom and Quality of Life Questionnaire (UFS- QoL )
* Safe access for the MRgFUS possible (anatomical position of the fibroids): Pelvic magnetic resonance imaging to document the number, location and size of fibroids and to exclude malignancy and other pelvic pathologies; necessary to determine whether MRgFUS can be performed technically (presence of a stable ultrasound window and exclusion of scars in the access path)
* ≤ 5 fibroids requiring treatment
* Fibroids with a diameter ≤ 10 cm
* Total myoma volume ≤ 400 ml
* Patient is suitable for treatment with MRgFUS-TUF as well as for myomectomy
* Desire for least invasive treatment
* Indication for hysteroscopy and fractionated abrasion depending on the bleeding pattern and endometrial thickness and structure have been critically tested in advance.
* inconspicuous cytological smear of the cervix uteri not older than 12 months
* No previous uterine surgery / intervention
* Female patients aged> 18 years. Patients of reproductive age must adhere to appropriate contraception until 6 months after the procedure. (Methods of contraception that meet the criteria of highly effective contraception in the sense of the Note for guidance on non- clinical safety studies for the conduct of human clinical trials for meet pharmaceuticals [CPMP / ICH / 286/95 mod ]). Patients of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* Karnofsky index ≥ 70
* Given medical operability
* Written consent of the patient

Exclusion Criteria:

* Pretreatment with ulipristal acetate ( Esmya ) ≤ 2 months
* Suspected Malignancy (absolute)
* Pregnancy (absolute)
* acute inflammatory process (absolute)
* Uterus myomatosis with more than 5 fibroids (relative, case-by-case decision)
* Uterine fibroids with a diameter over 10 cm (absolute)
* insufficient sound window can be reached for treatment (eg intestinal overlays, large scars in the acoustic window, very dorsal position of the fibroid)
* subserous stalked fibroids
* Inaccessible location of fibroids
* Scarring in the treatment area
* Recurring abortions
* general contraindications to MR contrast agents
* MRI contraindications
* Presence of pacemaker or metal implants
* Karnofsky Index <70
* Severe hepatic dysfunction (Aspartat-Aminotransferase (AST) / Transaminasen Alanin-Amino-transferase (ALT)> 3.5x ULN (upper limit of normal), Alkalische Phosphatase (AP)> 6xULN)
* Active CHD (congenital heart disease), (symptoms present), cardiomyopathy or heart failure in NYHA (New York Heart Association) and EF (ejection fraction) stage III-IV <45%
* Serious internistic side-diseases or an acute infection
* Chronic inflammatory bowel disease
* Pregnancy or lactation
* Participation in another interventional study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
WAI question 4 | Until at least three consecutive days questionnaire was answered as indicated, up to 12 months
  Time to sustainably return to normal activities, based on the daily Work Activity Index (WAI) dimension, "Estimated Impairment of Disease Performance". The return to normal activities is considered to be given if the question "Hindrance of medical condition or injury at work?" (min max: 1: 'in my opinion, I am completely unable to work', 6: 'No Disability') is answered for at least three consecutive days with "No Disability" (6) or "I can do my job, but have complaints" (5).
Symptom Severity Score of the UFS-QoL | 12 months after treatment
  The symptom severity is determined to be the co- primary endpoint for assessing therapeutic efficacy, based on the SSS (Symptom Severity Score) of the UFS-QoL (Uterine fibroid symptom and quality of life questionnaire). The co-primary assessment is performed 12 months after the primary treatment and for the evaluation the proportion of patients with at least 25 points improvement in the SSS is determined (0-100 scale, 100 indicating very strong symptoms, 0 no or low symptoms).

SECONDARY OUTCOMES:
Hospital stay in days | 12 months after treatment
Pain according to visual analog scale | 12 months after treatment
  Visual analog scale ranges from 0-100, 0 indicating no pain, 100 severe pain
Number of Adverse Events (AEs) | 12 months after treatment
Number of postinterventional/postsurgery treatment complications | 12 months after treatment
Number of re-interventions | 12 months after treatment
Alleviation of symptoms (irregular period, unfulfilled wish for child, pain, quality of life according to UFS-QoL | 12 months after treatment
  QoL: Quality of Life score regarding symptoms, ranges from 0-100, 0 indicating very low QoL, 100 indicating very high QoL
Health related quality of life according to UFS-QoL | 12 months after treatment
  QoL: Quality of Life score regarding health, ranges from 0-100, 0 indicating very low QoL, 100 indicating very high QoL
Sexuality related parameters according to UFS-QoL | 12 months after treatment
  QoL: Quality of Life score regarding sexuality, ranges from 0-100, 0 indicating very low QoL, 100 indicating very high QoL
Number of pregnancies and live births | 12 months after treatment
Number of late complications like venous thromboembolisms within Follow up time frame | 12 months after treatment
Number of fibroid recurrences (de novo fibroids) within Follow up time frame | 12 months after treatment
Time period until return to normal physical activities, measured by the rate of patients, who achieved an a priori clinically relevant reduction of SSS of UFS-QoL | 12 months after treatment
  at timepoints: months 1, 3 and 6 compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten O Götze, PD Dr. med., Principal Investigator — Krankenhaus Nordwest
Locations (4):
- Germany (4):
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - FOKUS Radiologische Gemeinschaftspraxis, Göttingen
  - Leipzig University, Leipzig
  - Marienhospital, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.aerzteblatt.de/nachrichten/98991/Erster-G-BA-Auftrag-zu...1%20von%202%2027.11.2018%2014:10